CLINICAL TRIAL: NCT04445168
Title: Intervention Based in Primary Care to Increase Physical Activity Among Inactive Adults With Prediabetes and Diabetes
Brief Title: Randomized Trial of Exercise Promotion in Primary Care
Acronym: EPPC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KPSC IRB#10106M
Record Dates: First submitted 2020-06-16; First posted 2020-06-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: PreDiabetes; Diabetes; Sedentary Behavior
Keywords: Physical activity; Randomized trial; Primary care
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants assigned to usual care may receive advice from their primary care physician to increase their physical activity. They will receive handouts about every 6 weeks on general health topics.
- Intervention (Experimental): Participants assigned to the intervention arm will receive telephone-based motivational interviews with trained interventionists to encourage increases in physical activity.
  Interventions: Behavioral: Telephone-based motivational interviews

INTERVENTIONS:
Behavioral: Telephone-based motivational interviews — 2-year telephone-based motivational interviews to increase physical activity.
  Arms: Intervention

SUMMARY:
Millions of Americans have diabetes or prediabetes, for which regular physical activity can reduce risks of unfavorable outcomes of these conditions. This study will test the effects of an evidence-based intervention in the primary care setting on increasing physical activity among these individuals. If effective, it can be broadly implemented in primary care.

ELIGIBILITY:
Inclusion Criteria:

Able to speak English or Spanish, Inactive defined as less than 30 minutes of MVPA per week, Prediabetes or diabetes not prescribed insulin, Kaiser Permanente member for at least 12 months, Receives primary care at the Fontana Medical Center, Body mass index between 18.5 and 40 kg/m2,

Exclusion Criteria:

Current use of insulin, Cardiovascular event in the past 6 months or other condition that limits physical activity, Pregnancy, breastfeeding or planning pregnancy in next 2 years, Current participation in another clinical trial or research study, Plans to move out of the area in next 2 years,

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Moderate to vigorous physical activity (MVPA) | 12 months
  Accelerometer-derived 7-day MVPA
Moderate to vigorous physical activity (MVPA) | 24 months
  Accelerometer-derived 7-day MVPA

SECONDARY OUTCOMES:
Weight | 12 months
  Weight assessed from electronic medical records
Weight | 24 months
  Weight assessed from electronic medical records
Systolic blood pressure | 12 months
  Systolic blood pressure assessed from electronic medical records
Systolic blood pressure | 24 months
  Systolic blood pressure assessed from electronic medical records
Diastolic blood pressure | 12 months
  Diastolic blood pressure assessed from electronic medical records
Diastolic blood pressure | 24 months
  Diastolic blood pressure assessed from electronic medical records
HbA1c | 12 months
  HbA1c assessed from electronic medical records
HbA1c | 24 months
  HbA1c assessed from electronic medical records
Health-related quality of life | 12 months
  Assessed from the short form (SF-8) instrument; scale 0 - 100, higher is more favorable quality of life
Health-related quality of life | 24 months
  Assessed from the short form-8 instrument; scale 0 - 100, higher is more favorable quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Southern California, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No